CLINICAL TRIAL: NCT05122767
Title: Safety, Tolerability and Drug-drug Interactions of Short-course Treatment of Latent Tuberculosis Infection With High-dose Once-weekly Rifapentine and Isoniazid (3HP) Among Infants, Children and Adolescents Living With HIV Taking Dolutegravir-based Antiretroviral Treatment
Brief Title: Rifapentine and Isoniazid TB Preventive Therapy (3HP) for Children Taking Dolutegravir-based Antiretroviral Treatment (DOLPHIN KIDS)
Acronym: DOLPHIN KIDS
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Aurum Institute NPC (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00280272
Record Dates: First submitted 2021-08-09; First posted 2021-11-17 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Tuberculosis; HIV
Keywords: TB; 3HP; pharmacokinetic; rifapentine; isoniazid; dolutegravir
MeSH Terms: conditions — Tuberculosis | interventions — dolutegravir

STUDY DESIGN:
Intervention Model Description: Single-arm, multi-center, Phase I/II clinical trial, in two groups. Individuals with HIV infection taking Efavirenz (EFV), nevirapine (NVP) or lopinavir/ritonavir (LPV/r) and two nucleoside reverse transcriptase inhibitors (NRTI) who have undetectable HIV viral load (< 50 copies/mL) and an indication for TPT, will be switched to DTG with tenofovir/emtricitabine (TDF/FTC), tenofovir/lamivudine (TDF/3TC), abacavir/lamivudine (ABC/3TC) or zidovudine/lamivudine (AZT/3TC) in accordance with South African National HIV Guidelines. Groups 1 and 2 will receive weekly HP for 12 total doses starting 4 weeks after initiating DTG. Individuals who are on an existing DTG-based plus two NRTI ART regimen for at least four weeks (and have not received efavirenz, or nevirapine or lopinavir/ritonavir for at least four weeks) who have an undetectable HIV viral load may also participate.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm in 4 groups (Experimental): There will be four groups. Group 1a and Group 1b will provide semi-intensive PK data and safety monitoring to allow for comparison of twice-daily dolutegravir exposures together with HP vs. when DTG is given alone. Group 2a and Group 2b will provide semi-intensive PK data and safety monitoring for either twice-daily or once-daily dolutegravir together with HIV vs when DTG is given alone. All groups will provide safety and tolerability data, HIV virologic outcome data, and information about dolutegravir and rifapentine PK.
  Interventions: Drug: Dolutegravir; Drug: 3HP

INTERVENTIONS:
Drug: Dolutegravir — Groups 1a/1b: Participants will take the FDA-approved weight-based DTG once daily + either TDF/FTC, TDF/3TC, ABC/3TC or AZT/3TC x 4 weeks. During HP treatment and for two weeks afterward, DTG dose will be increased to twice daily.
  Participants will continue with the NRTI regimen they have previously tolerated, except where their age and weight allow them to transition from either AZT or ABC to TDF, as per South African National ART Guidelines. HLA-B*5701 screening will therefore not be performed, as children will be currently taking and tolerating an ABC-containing regimen at enrolment. If any clinically suspected hypersensitivity reaction to ABC is suspected by history, ABC will not be continued.
  Groups 2a/2b: Participants will take weight-based DTG dosing twice or once daily, depending on the results of the modelled data for the Group 1a (for Group 2a) and/or Group 1b (for Group 2b) participants in the interim analysis.
Drug: 3HP — 3HP Dosing is by Age and Weight Children 2-15 years of age: 10-15kg (P 300mg, H 300mg); 16-23kg (P 450mg, H 500mg); 24-30kg (P 600mg, H 600mg); 31-34kg (P 750mg, H 700mg). Children 15-17 years, >=30kg (P 900mg, H 900mg)

SUMMARY:
Single-arm, multi-center, Phase I/II clinical trial, in two groups. Individuals with HIV infection taking Efavirenz (EFV), nevirapine (NVP) or lopinavir/ritonavir (LPV/r) and two nucleoside reverse transcriptase inhibitors (NRTI) who have undetectable HIV viral load (VL) (< 50 copies/mL) and an indication for tuberculosis (TB) preventive treatment (TPT), will be switched to dolutegravir (DTG) with tenofovir/emtricitabine (TDF/FTC), tenofovir/lamivudine (TDF/3TC), abacavir/lamivudine (ABC/3TC) or zidovudine/lamivudine (AZT/3TC) in accordance with South African National HIV Guidelines. Groups 1 and 2 will receive weekly HP for 12 total doses starting 4 weeks after initiating DTG. Individuals who are on an existing DTG-based plus two NRTI antiretroviral therapy (ART) regimen for at least four weeks (and have not received efavirenz, or nevirapine or lopinavir/ritonavir for at least four weeks) who have an undetectable HIV viral load may also participate.

DETAILED DESCRIPTION:
Group 1a (n=15): 15 participants aged 2-17 years of age will have suppressed viral load and take weight-based dosing of dolutegravir once daily with two nucleoside reverse transcriptase inhibitors (NRTIs) from Days 1-28. Semi-intensive pharmacokinetic (PK) sampling for dolutegravir will be performed on Day 28. Participants start twice-daily dolutegravir and will receive once-weekly rifapentine (RPT) and isoniazid (INH) (3HP) for 12 total doses beginning on Day 29. Semi-intensive PK sampling for dolutegravir will be performed on Day 46 (3 days after the 3rd dose of HP). Additional sparse PK sampling for dolutegravir (trough concentrations (CT)) will be performed on Days 44 and 48. Semi-intensive PK sampling for RPT will be performed on day 78. PK assessments will not be performed for isoniazid given that it's a well-studied drug in children. VL will be measured at baseline (week 0) and week 7 (after 3 doses of 3HP) and week 24 (8 weeks after the last dose of 3HP). Safety labs (complete blood count (CBC), urea and electrolytes (U&E), creatinine, and liver function tests (LFT)) will be obtained at baseline (week 0), and weeks 4, 7, 12, 16, 20, and 24.

Interim analysis will occur when all Group 1a participants have completed the 7-week semi-intensive PK visit (HP week 3). Enrolment into Group 2a (but not group 1b) will commence once this interim analysis is complete. Enrolment into group 1b will not be paused during this interim analysis. The interim analysis will assess PK, safety, and VL data. PK data will be modeled to assess the appropriateness of studying once-daily DTG dosing with co-administration of 3HP. The subsequent 30-45 participants age 2-17 years of age in Group 2a will receive twice or once-daily dosing of DTG, respectively, depending on PK modeling results.

Group 1b (n=8 ): All participants less than 2 years of age with a suppressed viral load will take weight-based dosing of dolutegravir once daily with two nucleoside reverse transcriptase inhibitors (NRTIs) from Days 1-28. Semi-intensive PK sampling for dolutegravir will be performed on Day 28. Participants start twice-daily dolutegravir and will receive once-weekly HP for 12 total doses beginning on Day 29. Semi-intensive PK sampling for dolutegravir will be performed on Day 46 (3 days after the 3rd dose of HP). Additional sparse PK sampling for dolutegravir (trough concentrations (CT)) will be performed on Days 44 and 48. Semi-intensive PK sampling for RPT will be performed on day 78. PK assessments will not be performed for isoniazid given that it's a well-studied drug in children. VL will be measured at baseline (week 0) and weeks 7 and 24. Safety labs (complete blood count (CBC), urea and electrolytes (U&E), creatinine, and liver function tests (LFT)) will be obtained at baseline (week 0), and weeks 4, 7, 12, 16, 20 and 24.

Interim analysis will occur when all Group 1b participants have completed the 7-week semi-intensive PK visit (HP week 3). Enrolment into group 2b (but not group 2a) will commence once this interim analysis is complete. Enrolment into group 2a will not be paused during this interim analysis. Interim analysis will assess PK, safety, and VL data. PK data will be modeled to assess the appropriateness of studying once-daily DTG dosing with co-administration of 3HP. The subsequent 16-24 participants in group 2b will receive twice or once-daily dosing of DTG, respectively, depending on population PK modeling results in this interim group.

Group 1b may or may not occur in parallel with Group 1a. This depends on the availability of dosing and a child-friendly formulation for 3HP in children 2 years and younger.

Group 2a (n=45 or 30): In the case where we proceed with evaluating once-daily DTG with 3HP in children 2-17 years of age, an additional 45 participants with suppressed viral load will be enrolled. In the case where we proceed with evaluating twice-daily DTG dosing with 3HP, an additional 30 participants with suppressed viral load will be enrolled. Both groups will take dolutegravir once daily from days 1-28 (weeks 1-4). On day 28, semi-intensive PK sampling for dolutegravir will be performed (prior to any HP dose). On day 29 (week 5), participants will either continue to take once daily DTG or their daily weight-based DTG dose will be increased to twice daily (based on group 1a data) and the first of the 12 HP weekly weight-based HP doses will be provided. Semi-intensive PK sampling for DTG will be performed on day 46 (2-4 days post third HP dose). Additional sparse PK sampling for dolutegravir (trough concentrations (CT)) will be performed on Days 44 and 48. Semi-intensive PK sampling for RPT will be performed on day 78. Viral load will be measured at baseline (screening, week 0) and at weeks 7 and 24. Safety labs (complete blood count (CBC), urea and electrolytes (U&E), and creatinine, and liver function tests (LFT)) will be obtained at baseline (screening, week 0), and weeks 4, 7, 12, 16, 20 and 24. Analysis will occur when 30 participants, in the case of twice daily DTG dosing, or 45 participants, in the case of once daily DTG dosing, have all completed the Week 24 visit.

Group 2a will occur following interim results from Group 1a, but may proceed without results from Group 1b.

Group 2b (n=24 or 16): In the case where we proceed with evaluating once daily DTG with 3HP in children less than 2 years of age, an additional 24 participants with suppressed viral load will be enrolled. In the case where we proceed with evaluating twice daily DTG dosing with 3HP, an additional 16 participants less than 2 years of age with suppressed viral load will be enrolled. Both groups would take dolutegravir once daily from days 1-28 (weeks 1-4). On day 28, semi-intensive PK sampling for dolutegravir will be performed (prior to any HP dose). On day 29 (week 5), participants will either continue to take once daily DTG or their daily weight-based DTG dose will be increased to twice daily (based on group 1a and group 1b data) and the first of the 12 HP weekly weight-based HP doses will be provided. Semi-intensive PK sampling for DTG will be performed on day 46 (3 days post third HP dose). Additional sparse PK sampling for dolutegravir (trough concentrations (CT)) will be performed on Days 44 and 48. Semi-intensive PK sampling for RPT will be performed on day 78. Viral load will be measured at baseline (screening, week 0) and at weeks 7 and 24. Safety labs (complete blood count (CBC), urea and electrolytes (U&E), and creatinine, and liver function tests (LFT)) will be obtained at baseline (screening, week 0), and weeks 4, 7, 12, 16, 20 and 24. Analysis will occur when 16 participants, in the case of twice-daily DTG dosing, or 24 participants, in the case of once-daily DTG dosing, have all completed the Week 24 visit.

Group 2b will follow Group 1b and may or may not occur in parallel with Group 2a. This depends on the availability of dosing and a child-friendly formulation for 3HP in children 2 years and younger.

ELIGIBILITY:
Inclusion criteria include:

* Age 3 months through 17 years
* Weight > 3 kg
* Documented HIV infection by DNA polymerase chain reaction (PCR) or plasma RNA-PCR if <18 months and by HIV-ELISA if 18 months and confirmed with a DNA PCR or RNA-PCR from an independent sample
* Undetectable HIV-1 viral load

Exclusion criteria

* Confirmed or suspected TB disease (evidenced by symptoms and/or clinical exam findings and/or chest radiographic findings suggestive of TB, positive mycobacterial culture or molecular TB testing, or currently on TB treatment for active TB disease)
* Likely to move from the study area during the study period
* Known exposure to TB cases with known or suspected resistance to isoniazid or rifampicin in the source case
* TB treatment within the past year
* Prior completion of a TPT course without re-exposure to persons with infectious TB since TPT completion
* Receipt of once-daily INH for >30 days that was given for at least 14 consecutive days in the 30 days prior to enrolment.
* Sensitivity or intolerance to dolutegravir, isoniazid, or rifamycins
* Suspected acute hepatitis or known chronic or unstable liver disease^; HBsAg positivity or anti-hepatitis A virus (HAV) Immunoglobulin M (IgM) antibody; any infant born to a Hepatitis C positive mother in whom in utero infection in the infant is unknown or under evaluation
* alanine aminotransferase (ALT) > 3 times the upper limit of normal (ULN)
* Total bilirubin > 2 .5 times the ULN
* Absolute neutrophil count (ANC) ≤ 750 cells/mm3
* Estimated creatinine clearance < 60 ml/min (Bedside Schwartz formula)*
* Pregnancy or breastfeeding (infant of a breastfeeding mother is allowed)
* Women of childbearing potential who are unable or unwilling to use two forms of contraception**
* Weight for age Z score below 2 or severe clinical malnutrition
* On prohibited medications e.g. dofetilide (see Appendix 1)
* Known porphyria

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2025-07-04 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
PK sampling of Dolutegravir - ka parameter | PK sampling at Week 4 (Day 29) and Week 7 (Days 44, 46, and 48) to be reported at end of trial
  Absorption rate constant (ka) in the presence or absence of once weekly HP (all groups)
PK sampling of Dolutegravir - Vd parameter | PK sampling at Week 4 (Day 29) and Week 7 (Days 44, 46, and 48) to be reported at end of trial
  Volume of distribution in the presence or absence of once weekly HP (all groups)
PK sampling of Dolutegravir - Cl/F parameter | PK sampling at Week 4 (Day 29) and Week 7 (Days 44, 46, and 48) to be reported at end of trial
  Oral clearance in the presence or absence of once weekly HP (all groups)
PK sampling of Dolutegravir - AUC parameter | PK sampling at Week 4 (Day 29) and Week 7 (Days 44, 46, and 48) to be reported at end of trial
  Area under the plasma drug concentration-time curve in the presence or absence of once weekly HP (all groups)
PK sampling of Dolutegravir - Ctau parameter | PK sampling at Week 4 (Day 29) and Week 7 (Days 44, 46, and 48) to be reported at end of trial
  Trough concentration in the presence or absence of once weekly HP (all groups)

SECONDARY OUTCOMES:
Adverse Events | Adverse events to be collected from Week 1 through Week 24, to be reported throughout the trial
  Grade 3 or higher adverse events (AE) (all groups)
HIV-1 RNA viral load | HIV viral load to be measured at Screening, and Weeks 7 and 24, to be reported at end of trial
  HIV-1 RNA viral load (copies/ml) (all groups)
PK sampling of RPT - AUC parameter | PK sampling at Week 12 (Day 78) to be reported at end of trial
  Area under curve (AUC) (all groups)
PK sampling of RPT - Cmax parameter | PK sampling at Week 12 (Day 78) to be reported at end of trial
  Maximum concentration (Cmax) (all groups)
PK sampling of RPT - Ctau parameter | PK sampling at Week 12 (Day 78) to be reported at end of trial
  Trough concentration (Ctau) (all groups)
DTG Dose selection | Dose selection will be determined at the interim analysis to be conducted when all participants in Groups 1a and 1b have completed the Week 7 PK visit. Based upon these results, Groups 2a and 2b will receive DTG either once or twice daily.
  Dose options for DTG with once-weekly HP derived by simulation using nonlinear mixed effects models

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Salazar-Austin, Principal Investigator — JHU SOM Ped Infectious Disease
Locations (2):
- South Africa (2):
  - The Aurum Institute: Pretoria Clinical Research Centre, Pretoria, Gauteng
  - Peri Natal HIV Research Unit - Klerksdorp Tshepong Hospital, Klerksdorp, North West

IPD SHARING:
Plan to Share IPD: No